CLINICAL TRIAL: NCT07126353
Title: Metabolic Risk Assessment in Prepubertal Children With Congenital Hypothyroidism (IpoMet)
Brief Title: Metabolic Risk Assessment in Prepubertal Children With Congenital Hypothyroidism
Acronym: IpoMet
Status: Not yet recruiting | Type: Observational
Sponsor: Buzzi Children's Hospital (Other)
Collaborators: Federico II University (Other); IRCCS Ospedale San Raffaele (Other); Policlinico di Bari Giovanni XXIII (Unknown); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other); Azienda Ospedaliera Sant'Anna (Other); University Hospital Perugia (Unknown); University of L'Aquila (Other); Clinica Pediatrica Università di Novara (Unknown); Santobono-Pausilpon Hospital (Unknown); Policlinico G . Martino, Messina Italy (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University Hospital of Ancona (Unknown)
Responsible Party: Principal Investigator, Valeria Calcaterra, Prof, Buzzi Children's Hospital
Other Study IDs: CET 503-2024
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Congenital Hypothyroidism; Metabolic Syndrome
Keywords: Congenital hypothyroidism; metabolic syndrome; Obesity
MeSH Terms: conditions — Congenital Hypothyroidism; Metabolic Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Permanent congenital hypothyroidism: 170 patients in prepubertal age.
  Interventions: Other: prospective observational study (clinical, hormonal and auxological data)
- Healthy childrens normal weight: 170 childrens in prepubertal age.
  Interventions: Other: prospective observational study (clinical, hormonal and auxological data)
- Healthy childrens overweight/obese: 170 patients in prepubertal age
  Interventions: Other: prospective observational study (clinical, hormonal and auxological data)

INTERVENTIONS:
Other: prospective observational study (clinical, hormonal and auxological data) — We collect clinical, hormonal and auxological data and compare them between the two groups.

SUMMARY:
We propose a multicenter prospective study to define the prevalence and severity score of metabolic syndrome in a prepubertal pediatric cohort with congenital hypothyroidism, compared to a healthy and normal-weight pediatric population. These data will help to define whether hypothyroidism can be considered a risk factor for the metabolic health of the pediatric population. The possible identification of an at-risk metabolic profile will provide useful information to optimize the diagnostic and monitoring pathway for affected children.

DETAILED DESCRIPTION:
Primary congenital hypothyroidism is the most common endocrine disorder in childhood and can present in either a permanent or transient form. Prolonged thyroid hormone deficiency can cause widespread damage affecting multiple organs and systems. Exposure to thyroid hormone deficiency during fetal and/or neonatal life has particularly severe consequences on the central nervous system, leading to neurocognitive delay. Appropriate and timely hormone replacement therapy (L-thyroxine) can prevent such outcomes, provided it is initiated early.

Thyroid hormones play a crucial role not only in growth and organ development but also in metabolic homeostasis. Thyroid function lies at the crossroads of multiple metabolic pathways. They have multiple effects on glucose and lipid metabolism, specifically by increasing glucose levels, fatty acid oxidation in muscle and liver, and lipolysis in adipose tissue. They also contribute to blood pressure regulation, thereby influencing the prevalence of metabolic syndrome, which is itself a key predictor of type 2 diabetes, cardiovascular diseases, and neurodegenerative conditions.Thyroid function plays a central regulatory role at the intersection of key metabolic pathways. Although, the role of thyroid hormones in metabolic processes is well established, and a bidirectional relationship between metabolic dysfunction and thyroid hypofunction has been reported in the adult population, data on metabolic risk in pediatric patients with congenital hypothyroidism are currently lacking.

The primary aim of this multicenter project is to assess the prevalence of metabolic syndrome in patients with congenital hypothyroidism and to determine whether this population presents a higher metabolic risk profile compared to the general population. As secondary objectives, this prospective study aims to:

1. Define the prevalence and severity score of metabolic syndrome in a prepubertal pediatric cohort with congenital hypothyroidism, compared to a pediatric population with obesity.
2. Evaluate the correlations between individual metabolic dysfunction parameters and the clinical and hormonal profile (including thyroid hormone levels and thyroid hormone sensitivity indices).
3. Assess the correlations between the metabolic profile and renal function.
4. Assess the correlations between the hormonal profile and renal function. To achieve these objectives, auxological parameters, vital signs (including blood pressure and heart rate), and metabolic profile data (glucose and lipid profiles, renal function, and hormonal status - FT3, FT4, TSH and thyroid hormone resistence indices TSHI, TT4RI, TT3RI, TFQI, PTFQI) will be collected for each enrolled subject. These parameters will be evaluated on peripheral blood samples collected during routine blood monitoring already scheduled according to established follow up. The potential presence of metabolic syndrome will be evaluated in each enrolled patient. The severity of the metabolic disorder will be evaluated using the Metabolic Score (MetS).

Data analysis will be performed using the statistical packages R 4.0.5 (R Core Team, 2021) and STATA (version 15.1, 2017, Stata Corporation, College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Pubertal stage Tanner 1
* Permanent congenital hypothyroidism
* All ethnic groups
* Informed consent signature

Exclusion Criteria:

* Age< 5 years
* Pubertal stage Tanner 2-5
* Transient congenital hypothyroidism or other type of hypothyroidism

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We enrolled patients affected by permanent congenital hypothyroidism in prepubertal age and healthy childrens in prepubertal age to compare them with each other.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome (MS) | At the time of enrollment
  Presence of at least 3 of the following parameters:
  1. BMI z-score ≥ 2 and/or waist-to-height ratio (WHtR) > 0.5
  2. Fasting blood glucose ≥ 100 mg/dL and/or TryG index ≥ 7.88
  3. Total cholesterol ≥ 200 mg/dL
  4. HDL cholesterol < 40 mg/dL and/or LDL cholesterol ≥ 130 mg/dL
  5. Triglycerides (TG) ≥ 100 mg/dL for ages 0-9 years; ≥ 130 mg/dL for ages >10 years
  6. Systolic and/or diastolic blood pressure (SBP and/or DBP) ≥ 90th percentile for age and sex
Metabolic score (MeTs) | At the time of enrollment
  Males MetS z-score = -4.931 + 0.2804 * BMI z-score - 0.0257 * HDL + 0.0189 * SBP + 0.6240 * log(triglycerides) + 0.0140 * fasting glucose
  Females MetS z-score = -4.3757 + 0.4849 * BMI z-score - 0.0176 * HDL-C + 0.0257 * SBP + 0.3172 * log(triglycerides) + 0.0083 * fasting glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jostel A, Ryder WD, Shalet SM. The use of thyroid function tests in the diagnosis of hypopituitarism: definition and evaluation of the TSH Index. Clin Endocrinol (Oxf). 2009 Oct;71(4):529-34. doi: 10.1111/j.1365-2265.2009.03534.x. Epub 2009 Feb 18. PMID 19226261
- [Background] Iwamoto Y, Kimura T, Tatsumi F, Sugisaki T, Kubo M, Nakao E, Dan K, Wamata R, Iwamoto H, Takahashi K, Sanada J, Fushimi Y, Katakura Y, Shimoda M, Nakanishi S, Mune T, Kaku K, Kaneto H. Effect of Hyperglycemia-Related Acute Metabolic Disturbance on Thyroid Function Parameters in Adults. Front Endocrinol (Lausanne). 2022 May 12;13:869869. doi: 10.3389/fendo.2022.869869. eCollection 2022. PMID 35634497
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554
- [Background] Laclaustra M, Moreno-Franco B, Lou-Bonafonte JM, Mateo-Gallego R, Casasnovas JA, Guallar-Castillon P, Cenarro A, Civeira F. Impaired Sensitivity to Thyroid Hormones Is Associated With Diabetes and Metabolic Syndrome. Diabetes Care. 2019 Feb;42(2):303-310. doi: 10.2337/dc18-1410. Epub 2018 Dec 14. PMID 30552134
- [Background] Lakhani G, Patel P, Patel TC. A Cross-Sectional Study on the Prevalence of Subclinical Hypothyroidism in Metabolic Syndrome Patients at a Tertiary Care Hospital. Cureus. 2024 Aug 26;16(8):e67851. doi: 10.7759/cureus.67851. eCollection 2024 Aug. PMID 39323691
- [Background] Thakur R, Kumar S, Neeraj RK, Saleem M, Kumar C, Mohan L. Evaluation of the Association between Insulin Resistance and Subclinical Hypothyroidism Using Triglyceride-Glucose Index: a Cross-Sectional Study. Maedica (Bucur). 2024 Jun;19(2):255-259. doi: 10.26574/maedica.2024.19.2.255. PMID 39188835
- [Background] Verma DP, Chaudhary SC, Singh A, Sawlani KK, Gupta KK, Usman K, Reddy HD, Patel ML, Verma SK, Atam V. Hypothyroidism in Metabolic Syndrome. Ann Afr Med. 2024 Oct 1;23(4):717-722. doi: 10.4103/aam.aam_25_24. Epub 2024 Sep 14. PMID 39279179
- [Background] Xie H, Li N, Zhou G, He Z, Xu X, Liu Q, Wang H, Han J, Shen L, Yu P, Chen J, Chen X. The association between the thyroid feedback quantile-based index and serum uric acid in U.S. adults. Eur J Med Res. 2023 Jul 27;28(1):259. doi: 10.1186/s40001-023-01214-3. PMID 37501165
- [Background] Xie Y, Wang Z, Chen Z. Analysis of Subclinical Thyroid Dysfunction and Metabolic Abnormality in 28568 Healthy People. Int J Endocrinol. 2023 Oct 16;2023:5216945. doi: 10.1155/2023/5216945. eCollection 2023. PMID 37876378
- [Background] Zhong L, Liu S, Yang Y, Xie T, Liu J, Zhao H, Tan G. Metabolic syndrome and risk of subclinical hypothyroidism: a systematic review and meta-analysis. Front Endocrinol (Lausanne). 2024 Jun 25;15:1399236. doi: 10.3389/fendo.2024.1399236. eCollection 2024. PMID 38982986
- [Background] Di Bonito P, Corica D, Marzuillo P, Di Sessa A, Licenziati MR, Faienza MF, Calcaterra V, Franco F, Maltoni G, Valerio G, Wasniewska M. Sensitivity to Thyroid Hormones and Reduced Glomerular Filtration in Children and Adolescents with Overweight or Obesity. Horm Res Paediatr. 2024;97(4):383-387. doi: 10.1159/000534472. Epub 2023 Oct 9. PMID 37812927
- [Background] Calcaterra V, Mameli C, Macedoni M, De Silvestri A, Sgambetterra L, Nosenzo F, Redaelli FC, Petitti A, Bosetti A, Zuccotti G. Investigating the connection among thyroid function, sensitivity to thyroid hormones, and metabolic syndrome in euthyroid children and adolescents affected by type 1 diabetes. J Pediatr Endocrinol Metab. 2024 Mar 12;37(4):347-352. doi: 10.1515/jpem-2023-0565. Print 2024 Apr 25. PMID 38462926
- [Background] Calcaterra V, Gazzarri A, De Silvestri A, Madia C, Baldassarre P, Rossi V, Garella V, Zuccotti G. Thyroid function, sensitivity to thyroid hormones, and metabolic syndrome in euthyroid children and adolescents with Down syndrome. J Endocrinol Invest. 2023 Nov;46(11):2319-2325. doi: 10.1007/s40618-023-02086-4. Epub 2023 Apr 11. PMID 37040064
- [Background] Biondi B. Subclinical Hypothyroidism in Patients with Obesity and Metabolic Syndrome: A Narrative Review. Nutrients. 2023 Dec 27;16(1):87. doi: 10.3390/nu16010087. PMID 38201918
- [Background] Alwan H, Ribero VA, Efthimiou O, Del Giovane C, Rodondi N, Duntas L. A systematic review and meta-analysis investigating the relationship between metabolic syndrome and the incidence of thyroid diseases. Endocrine. 2024 May;84(2):320-327. doi: 10.1007/s12020-023-03503-7. Epub 2023 Sep 9. PMID 37688711
- [Background] Alsulami SS, Baig M, Albeladi AH, Alyoubi SB, Alsubaie SA, Albeladi SA, Ghamri KA, Alraiqi AMS, Alyoubi SM, Almutairi WA. Correlation between Subclinical Hypothyroidism and Metabolic Syndrome: A Retrospective Study. Saudi J Med Med Sci. 2023 Jul-Sep;11(3):250-256. doi: 10.4103/sjmms.sjmms_225_22. Epub 2023 Jul 15. PMID 37533656
- [Background] Abha P, Keshari JR, Sinha SR, Nishant K, Kumari R, Prakash P. Association of Thyroid Function With Lipid Profile in Patients With Metabolic Syndrome: A Prospective Cross-Sectional Study in the Indian Population. Cureus. 2023 Sep 5;15(9):e44745. doi: 10.7759/cureus.44745. eCollection 2023 Sep. PMID 37809190